CLINICAL TRIAL: NCT03363529
Title: ROOM-LIGHT: Dynamic LED-light as Treatment for Depressed Patients in Inpatient Wards: A Feasibility Trial
Brief Title: ROOM-LIGHT: Dynamic LED-light as Treatment for Depressed Patients in Inpatient Wards
Acronym: ROOM-LIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Department of Photonics Engineering (Unknown); Chromaviso A/S (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ROOMLIGHT
Record Dates: First submitted 2017-11-16; First posted 2017-12-06 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Depression; Light; Therapy, Complications; Sleep Disorders, Circadian Rhythm
Keywords: Dynamic lighting, ipRGC
MeSH Terms: conditions — Depression; Sleep Disorders, Circadian Rhythm | interventions — Dynamic Light Scattering; Reference Standards

STUDY DESIGN:
Intervention Model Description: Standard versus dynamic lighting
Who Masked: Outcomes Assessor
Masking Description: Hamilton depression interview is done by external assessor blinded to condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Placebo Comparator): This study arm utilizes a standard lighting condition in the patient room
  Interventions: Device: Standard
- Dynamic (Experimental): This study arm utilizes a dynamic lighting from special designed lightfixtures in the ceiling and window sill.
  Interventions: Device: Dynamic light

INTERVENTIONS:
Device: Dynamic light — Dynamic lighting is light that changes in intensity and spectral distribution during the day
  Arms: Dynamic
Device: Standard — Standard lighting is non-dynamical light corresponding to standard hospital lighting.
  Arms: Standard

SUMMARY:
Depression is a major health challenge, and despite developments in pharmacotherapy and psychotherapy a substantial part of patients will only recover very slowly and incompletely, and 10-25 % of the patients are resistant to treatment. Therefore, new treatment initiatives are in demand. Chronotherapeutics can regulate diurnal rhythms and sleep, and have shown promising results on antidepressant effects. Among chronotherapeutic treatment modalities, Bright Light Therapy (BLT) has been used in treatment of depression and sleep disorders for several decades with both an antidepressant and a sleep improving effect. BLT has also been shown to augment antidepressant therapy.

Objectives. The objective of this trial is to investigate the feasibility of a combination of LED-light armatures aiming to mimic sunlight, when installed in the patient rooms of a psychiatric inpatient Ward. Investigators has opted for using a randomized design that will subsequently be tested in a larger clinical trial with depression severity as the primary outcome. In this feasibility study investigators will register the stability of the system, the influence of the light on patients regarding tolerability, comfort, depression level, and sleep. Investigators also so want to measure and collect specific light-data on the Non-image-forming light (NIF) by using specially designed light sensors to capture the spectral distribution of the light. Finally investigators will test the electronic case report form (eCRF) that has been designed for the trial.

Design. The design is a randomised controlled feasibility trial with two arms: an active dynamic light trial arm and a standard light trial arm with blinding of depression outcome assessors (Hamilton depression rating scale), data collection, and data analyses. Randomization will be with a rate for active and standard of 2 to 1.

DETAILED DESCRIPTION:
Inclusion and exclusion criteria. Inclusion: Major depression disorder, age > 18 years, informed consent and Danish speaking.

Exclusion: Severe suicidality, actual psychotic state, bipolar disorder and if the patient is subject to coercive measures of any kind.

Name and description of experimental and control intervention. The experimental intervention is the implementation of a dynamic LED-light system in two patient rooms. The system includes three elements: a window jamb built-in light panel, two ceiling mounted lamps, and a wall mounted lamp. All lamps will have a dynamic, time dependent frequency distribution and intensity of light. The control intervention is constant standard LED-light with two elements: two ceiling mounted lamps and a wall mounted lamp.

Primary and secondary outcomes.

Primary outcome:

1. Rate of patients discontinuing the trial due to discomfort from the lighting condition.

Secondary outcomes:

1. Mean scores on the visual comfort scale in the intervention period
2. Reduction in HAM-D17 scores from baseline to week 4 Trial size. In total 15 patients. All regulatory approvals has been met from the Danish Data Protection Agency, the regional Ethics Committee Agency, and the Mental Health Services of Copenhagen.

Time schedule. The first participant is expected to be enrolled in December 2017. The expected last follow-up of the last participant will be June 2018. Data will be analysed from June 2018 till December 2018. Manuscripts will be prepared from June 2017 and we expect to submit first manuscript January 2019.

ELIGIBILITY:
Inclusion Criteria:

* Major depression disorder
* Age > 18 years
* Informed consent and Danish speaking.

Exclusion Criteria:

* Severe suicidality
* Actual psychotic state
* Bipolar disorder
* Patient is subject to coercive measures of any kind.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Difference in numbers of drop out in the two groups | Week 4
  Number of patients in the two groups that drop out due to the standard or experimental lighting condition

SECONDARY OUTCOMES:
Visual comfort questionaire | Week 4
  Difference in scores in the Visual comfort questionaire
Change of depression level from baseline to endpoint | Change scores from baseline to week 4
  Difference in change scores on the Hamilton Depression Rating scale 17 item from baseline to week 4 in the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Martiny, DMSc, PhD, Principal Investigator — Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Locations (1):
- Mental Health Centre Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Volf C, Aggestrup AS, Svendsen SD, Hansen TS, Petersen PM, Dam-Hansen C, Knorr U, Petersen EE, Engstrom J, Hageman I, Jakobsen JC, Martiny K. Dynamic LED light versus static LED light for depressed inpatients: results from a randomized feasibility trial. Pilot Feasibility Stud. 2020 Jan 15;6:5. doi: 10.1186/s40814-019-0548-9. eCollection 2020. PMID 31956421